CLINICAL TRIAL: NCT05011669
Title: The Safety and Efficacy of Lurasidone With Different Initiation Dose in Chinese Acute Phase Patients With Schizophrenia: A Multi-Center, Prospective, Open-Label Study for 6 Weeks
Brief Title: The Safety and Efficacy of Lurasidone With Different Initiation Dose in Chinese Acute Phase Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSPCLAT-003
Record Dates: First submitted 2021-08-07; First posted 2021-08-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latuda® 40mg/d (Experimental)
  Interventions: Drug: Lurasidone
- Latuda® 80mg/d (Experimental)
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Oral administration with a meal or within 30 min after eating in the evening. The dosage could be adjusted from Day 8.

SUMMARY:
To evaluate the safety and efficacy of Lurasidone initiated with 40mg and 80mg in treatment with acute phase patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Subjects meet ICD10 criteria for a primary diagnosis of schizophrenia;
* Subjects have a score ≥ 4 on the CGI-S at Screening and Baseline;
* Subjects have a PANSS total score ≥ 70 and ≤ 120 at Screening and Baseline, with a score 4 (moderate) or higher in 2 or more items on the following PANSS items: delusions, conceptual disorganization, hallucinations, unusual thought content and suspiciousness;
* Subjects with acute (including recurrence /relapse and first episode) phase patients with schizophrenia;
* Ability to understand the contents of interview and provide written informed consent (If subject is unable to sign, subject's legal guardian or impartial witness shall sign the informed consent).

Exclusion Criteria:

* Subjects with severe or unstable physical diseases (including but not limited to severe or unstable cardiovascular diseases, cerebrovascular diseases, liver and kidney diseases) determined by the investigators;
* Subjects had a history of stomach or intestinal surgery or any other condition that could interfere with absorption, distribution, metabolism, or excretion of medications;
* Based on the judgement of investigators, subject has a history of refractory psychosis and/or subject has been treated with clozapine (for any reason) within 4 months of baseline;
* Subjects has used long-term antipsychotic drugs, e.g. Haloperidol decanoate injection, Fluphenazine decanoate injection, Risperidone microspheres injection, Paliperidone palmitate injection, Paliperidone palmitate injection (3M), in the following time prior to the enrolment;
* Subjects is at risk of suicide or self-mutilation behaviours or the act of endangering others, or other corresponding characteristic behaviour, or a history of suicide;
* Female subjects were pregnant (positive pregnancy test at screening) or breast-feeding or planning pregnancy for the duration of the study, or the partners of male subjects were planning pregnancy for the duration of the study;
* Need to use of disallowed concomitant therapy which is specified in the protocol;
* History of severe allergy or hypersensitivity;
* Currently has severe liver function impairment, or serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥3 times the upper limit of normal value;
* Creatinine clearance rate < 50mL/min Creatinine clearance rate*100%= Male: (140 - Age) x Weight(kg)/Serum creatinine (mg/dL) x 72 Female: 0.85*(140 - Age) x Weight(kg)/Serum creatinine (mg/dL) x 72
* A history of malignant tumors (including benign pituitary tumors);
* Any chronic organic disease of the central nervous system (excluding schizophrenia), such as CNS related tumors and inflammation, active seizures, vascular disease, Parkinson's disease, Alzheimer's disease, or other forms of dementia, myasthenia gravis, and other degenerative diseases. A history of mental retardation or persistent neurological symptoms caused by severe head injury;
* Subjects received electroconvulsive therapy (ECT) within 90 days prior to screening, or were expected to require ECT during the study;
* A history of neuroleptic malignant syndrome;
* Severe tardive dyskinesia, severe dystonia, or any other severe dyskinesia;
* Angioedema occurred after previous administration of lurasidone;
* The subject is participating in or has participated in other clinical trials, including the use of commercially available drugs or medical devices, within 30 days prior to the signing of the informed consent;
* Patients who had previously participated in a clinical study of lurasidone;
* Any other conditions judged by the investigators that not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Percentage of discontinuation due to adverse events | during the 6 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hospital, Beijing, Beijing Municipality, China